CLINICAL TRIAL: NCT04007575
Title: Magnetic Resonance CholangioPancreatography Signs for the Diagnosis of Caroli Disease
Brief Title: Study of New Imaging Criteria for the Diagnosis of Caroli's Disease
Acronym: IMACA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190470
Record Dates: First submitted 2019-06-04; First posted 2019-07-05 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Caroli Disease; Magnetic Resonance Imaging; Cholangiopancreatography
MeSH Terms: conditions — Caroli Disease | interventions — Cholangiopancreatography, Magnetic Resonance; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance CholangioPancreatography — The imaging data will be collected from the hospital records and image archiving system of the radiology departments of the University Hospitals
  Other Names: Magnetic Resonance Imaging

SUMMARY:
The Caroli disease is a very rare pathology that can be revealed early in childhood or in adulthood, whose diagnosis is based on Magnetic Resonance CholangioPancreatography, which shows the communication of these malformations with the rest of the biliary tree and allows to eliminate biliary stenosis. The radiologist has a central role in the diagnostic orientation between malformative intra-hepatic bile duct dilatation and obstructive benign or malignant intra-hepatic bile duct dilatation dilatation. However, imaging of Caroli disease is polymorphous and therefore subject to misinterpretation. The benefit of this research is to reduce diagnostic errors by highlighting imaging criteria specific to the Caroli disease

DETAILED DESCRIPTION:
The Magnetic Resonance CholangioPancreatography will have been performed in all patients using different Magnetic Resonance Imaging systems (Gyroscan Intera, Philips Medical Systems, Best in the Netherlands, Magnetom Avanto, Siemens Medical Solutions, and Signa Hdxt, General Electric Medical Systems) with a free-breathing three-dimensional high-spatial-resolution Fast Spin Echo sequence and/or a breath-hold two-dimensional single-shot sequence. Magnetic Resonance CholangioPancreatography may also include a Fast Spin Echo weighted T2-weighted sequence with fat-spectral saturation, a T1-weighted breath-suppressed gradient echo pulse sequence and a chemical shift sequence in phase and opposite phase, in the axial plane, and a weighted three-dimensional T1 saturated fat sequence after intravenous administration of gadolinium chelate. Images will be analyzed in consensus by two abdominal radiologists on a Picture Archiving and Communication System station and compared with the pathological results.

ELIGIBILITY:
Inclusion Criteria:

* were patients identified in the database of the hospitals who underwent
* a diagnosis of Caroli disease on an imaging report with bile duct dilatation limited to the intrahepatic biliary tree and
* an available Magnetic Resonance CholangioPancreatography on a Picture Archiving and Communication System.

Exclusion Criteria:

* obstructive benign or malignant proximal biliary stricture on Magnetic Resonance CholangioPancreatography
* prior surgical interventions for hepatobiliary disease except cholecystectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with illness or Caroli syndrome
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Intra-hepatic bile duct dilatation | 2 years
  study of intra-hepatic bile duct shape (qualitative measurement)
Intra-hepatic bile duct dilatation | 2 years
  intra-hepatic bile duct localisation (qualitative measurement)
Intra-hepatic bile duct dilatation | 2 years
  biliary calculi (qualitative measurement)
Intra-hepatic bile duct dilatation | 2 years
  dot sign (qualitative measurement)
Intra-hepatic bile duct dilatation | 2 years
  liver abnormalities (qualitative measurement)
Intra-hepatic bile duct dilatation | 2 years
  signs of portal hypertension (qualitative measurement)

SECONDARY OUTCOMES:
Pathological examination | 2 years
  Absence or presence of tumors
Pathological examination | 2 years
  Absence or presence of calculi
Biology | 2 years
  bilirubin level
Biology | 2 years
  Alkaline phosphatase level
Biology | 2 years
  Creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: LEWIN MAITE, MD, PhD, Principal Investigator — Paul Brousse hospital
Locations (1):
- Maite Lewin, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No